CLINICAL TRIAL: NCT02744677
Title: COngenital Multicenter Trial of Pulmonic vAlve Dysfunction Studying the SAPIEN 3 interventIONal THV
Brief Title: COMPASSION S3 - Evaluation of the SAPIEN 3 Transcatheter Heart Valve in Patients With Pulmonary Valve Dysfunction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-01
Record Dates: First submitted 2016-04-12; First posted 2016-04-20 (Estimated); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Complex Congenital Heart Defect; Dysfunctional RVOT Conduit; Pulmonary Valve Insufficiency; Pulmonary Valve Degeneration
Keywords: Tetralogy of Fallot; Aortic Valve Defect/Disease Resulting in Ross Procedure; Pulmonary Atresia; Pulmonary Stenosis; Truncus Arteriosus; Transposition of the Great Arteries; Transcatheter pulmonary valve implantation; Transcatheter pulmonary valve replacement; TPV; TPVR; TPVI
MeSH Terms: conditions — Pulmonary Valve Insufficiency; Tetralogy of Fallot; Aortic Valve Disease; Pulmonary Atresia; Pulmonary Valve Stenosis; Truncus Arteriosus, Persistent; Transposition of Great Vessels

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- TPVR - Main Cohort (Experimental): Subjects with a dysfunctional RVOT conduit or previously implanted surgical valve in the pulmonic position will undergo transcatheter pulmonary valve replacement (TPVR).
  Interventions: Device: SAPIEN 3 THV
- TPVR - THV Registry (Experimental): Subjects with a previously implanted transcatheter valve in the pulmonic position will undergo TPVR.
  Interventions: Device: SAPIEN 3/SAPIEN 3 Ultra RESILIA THV
- TPVR- S3UR Registry (Experimental): Subjects with a dysfunctional RVOT conduit or previously implanted surgical valve in the pulmonic position will undergo transcatheter pulmonary valve replacement (TPVR).
  Interventions: Device: SAPIEN 3 Ultra RESILIA THV

INTERVENTIONS:
Device: SAPIEN 3/SAPIEN 3 Ultra RESILIA THV — SAPIEN 3/SAPIEN 3 Ultra RESILIA THV in the pulmonic position
  Arms: TPVR - THV Registry
Device: SAPIEN 3 THV — SAPIEN 3 THV in the pulmonic position
  Arms: TPVR - Main Cohort
Device: SAPIEN 3 Ultra RESILIA THV — SAPIEN 3 Ultra RESILIA THV in the pulmonic position
  Arms: TPVR- S3UR Registry

SUMMARY:
This study will demonstrate the safety and effectiveness of the Edwards Lifesciences SAPIEN 3/SAPIEN 3 Ultra RESILIA Transcatheter Heart Valve (THV) Systems in subjects with a dysfunctional right ventricular outflow tract (RVOT) conduit or previously implanted valve in the pulmonic position with a clinical indication for intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Weight ≥ 20 kg (44 lbs.)
2. Dysfunctional RVOT conduit or previously implanted valve in the pulmonic position with a clinical indication for intervention and with a landing zone diameter ≥ 16.5 mm and ≤ 29 mm immediately prior to study device insertion as per the Instructions for Use
3. Subject presents with at least moderate PR and/or mean RVOT gradient ≥ 35 mmHg.
4. The subject/subject's legally authorized representative has been informed of the nature of the study, agrees to its provisions and has provided written informed consent.

Exclusion Criteria:

1. Active infection requiring current antibiotic therapy (if temporary illness, subject may be a candidate 2 weeks after discontinuation of antibiotics)
2. History of or active endocarditis (active treatment with antibiotics) within the past 180 days
3. Leukopenia, anemia, thrombocytopenia or any known blood clotting disorder
4. Inappropriate anatomy for femoral introduction and delivery of the study valve
5. Need for concomitant atrial septal defect or ventricular septal defect closure or other concomitant interventional procedures other than pulmonary artery or branch pulmonary artery stenting or angioplasty
6. Angiographic evidence of coronary artery compression that would result from transcatheter pulmonic valve implantation (TPVI)
7. Interventional/surgical procedures within 30 days prior to the TPVI procedure.
8. Any planned surgical, percutaneous coronary or peripheral procedure to be performed within the 30 day follow-up from the TPVI procedure.
9. History of or current intravenous drug use
10. Major or progressive non-cardiac disease resulting in a life expectancy of less than one year
11. Known hypersensitivity to aspirin or heparin and cannot be treated with other antiplatelet and/or antithrombotic medications
12. Known hypersensitivity to cobalt-chromium, nickel or contrast media that cannot be adequately premedicated
13. Participating in another investigational drug or device study that has not reached its primary endpoint.
14. Female who is lactating or pregnant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2016-07-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
THV dysfunction | 1 year
  Defined as a non-hierarchical composite of: RVOT reintervention, Moderate or greater total pulmonary regurgitation (PR) via Transthoracic Echocardiography (TTE), Mean RVOT gradient > 40 mmHg via TTE

SECONDARY OUTCOMES:
Device Success | Discharge, expected to be within 1-5 days post-procedure
  Defined as a composite of: 1) Single THV implanted in the desired location, 2) RV-PA peak-to-peak gradient < 35 mmHg post-implantation, 3) Less than moderate PR by discharge TTE (or earliest evaluable TTE), 4) Free of explant at 24 hours post-implantation.
Mean RVOT gradient | 6 months
Paravalvular and total PR | 6 months
RVOT reintervention | 6 months
Coronary artery compression requiring intervention | 30 days
Major vascular complications | 30 days
Life-threatening or disabling bleeding | 30 days
THV frame fracture | 6 months
Device-related endocarditis | 1 year
Death (all-cause, procedural and device-related) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: D. Scott Lim, MD, Principal Investigator — University of Virginia Medical Center; Vasilis Babaliaros, MD, Principal Investigator — Emory University Hospitals
Locations (25):
- United States (25):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of California, Los Angeles, Los Angeles, California
  - University of California,, San Francisco (UCSF), San Francisco, California
  - Childrens Hospital of Colorado, Aurora, Colorado
  - Emory University/Children's Healthcare of Atlanta, Atlanta, Georgia
  - University of Kentucky, Lexington, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - Mayo Clinic Rochester, Rochester, Minnesota
  - St. Louis Children's Hospital, St Louis, Missouri
  - Washington University Barnes- Jewish Medical/ St. Louis Children's Hospital, St Louis, Missouri
  - Columbia University Medical Center/NYPH, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - The Lindner Research Center at Christ Hospital, Cincinnati, Ohio
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Penn Presbyterian Medical Center, University of Pennsylvania/ Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - LeBonheur Children's Hopsital, Memphis, Tennessee
  - Medical City Dallas, Dallas, Texas
  - Children's Health System of Texas / UT Southwestern Medical Center, Dallas, Texas
  - Methodist San Antonio, San Antonio, Texas
  - Intermountain Heart Institute (IMC), Murray, Utah
  - University of Virginia (UVA), Charlottesville, Virginia
  - University of Washington/Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lim DS, Kim D, Aboulhosn J, Levi D, Fleming G, Hainstock M, Sommer R, Torres AJ, Zhao Y, Shirali G, Babaliaros V. Congenital Pulmonic Valve Dysfunction Treated With SAPIEN 3 Transcatheter Heart Valve (from the COMPASSION S3 Trial). Am J Cardiol. 2023 Mar 1;190:102-109. doi: 10.1016/j.amjcard.2022.12.010. Epub 2023 Jan 4. PMID 36608435